CLINICAL TRIAL: NCT01991522
Title: A Comprehensive Simulation-based Curriculum as a Means to Enhance Technical and Non-technical Skills in Colonoscopy: a Randomized Control Trial
Brief Title: A Randomized Control Trial of a Simulation-based Curriculum to Enhance Skills in Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Samir Grover, Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 13-197c
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curriculum Group (Experimental): The curriculum group will undergo a comprehensive curriculum in colonoscopy utilizing a virtual reality (VR) colonoscopic simulator. This curriculum involves 6 hours of interactive, small-group didactic teaching on colonoscopy interlaced with 8 hours of supervised one-on-one endoscopy VR simulation training with experienced endoscopists.
  Interventions: Behavioral: Curriculum Group
- Self-directed learning group (Active Comparator): The self-directed group will receive 8 hours of colonoscopic virtual reality (VR) simulation practice with an experienced endoscopist present, but without structured training.
  Interventions: Behavioral: Self-directed learning group

INTERVENTIONS:
Behavioral: Curriculum Group
  Arms: Curriculum Group
Behavioral: Self-directed learning group
  Arms: Self-directed learning group

SUMMARY:
Colonoscopy is a commonly used medical procedure. Medical and surgical residents learning colonoscopy typically learn the procedure experientially but simulation based teaching is increasingly being integrated into training programs. The optimal manner to teach colonoscopy on virtual-reality simulators is uncertain. We aim to test a curriculum in simulation-based colonoscopy with self-directed learning on simulators.

ELIGIBILITY:
Inclusion Criteria:

* Trainee endoscopists from the gastroenterology and general surgery programs at the University of Toronto

Exclusion Criteria:

* Greater than 20 colonoscopies performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir C Grover, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grover SC, Garg A, Scaffidi MA, Yu JJ, Plener IS, Yong E, Cino M, Grantcharov TP, Walsh CM. Impact of a simulation training curriculum on technical and nontechnical skills in colonoscopy: a randomized trial. Gastrointest Endosc. 2015 Dec;82(6):1072-9. doi: 10.1016/j.gie.2015.04.008. Epub 2015 May 23. PMID 26007221

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Curriculum Group | Self-directed Learning Group
Started | 16 | 17
Completed | 16 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curriculum Group | Self-directed Learning Group | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (1.3) | 29.7 (3.8) | 29.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 7 | 13 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Training program (gastroenterology, general surgery, or internal medicine) [Count of Participants; unit: Participants]
  Gastroenterology | 8 | 4 | 12
  General surgery | 8 | 11 | 19
  Internal Medicine | 0 | 2 | 2
Number of independent colonoscopies performed [Mean (Standard Deviation); unit: colonoscopies] | 0.6 (2.5) | 0.7 (2.9) | 0.65 (2.7)
Number of assisted colonoscopies performed [Mean (Standard Deviation); unit: Colonoscopies] | 2.7 (7.7) | 0.8 (1.5) | 1.7 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Transfer of Skills to Clinical Colonoscopy
Description: The Joint Advisory Group (JAG) Direct Observation of Procedural Skills (DOPS) tool is a tool to assess colonoscopic competency and includes ratings of the following domains: (i) assessment, consent and communication; (ii) safety and sedation; (iii) endoscopic skills during insertion and withdrawal; and, (iv) diagnostic and therapeutic ability. Scores range from 0-100, with higher scores representing higher colonoscopic competency. These were measured across two endoscopic procedures, performed consecutively within two weeks of completion of the course. Data from two procedures were used to limit the influence of spurious findings from single procedures.
Time Frame: less than 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curriculum Group | Self-directed Learning Group
Number analyzed (Participants) | 16 | 17
units on a scale
  Procedure 1 | 72.2 (10.9) | 31.8 (14.8)
  Procedure 2 | 71.9 (16.7) | 32.3 (18.3)

2. Secondary Outcome: Retention of Clinical Skills
Description: The Joint Advisory Group (JAG) Direct Observation of Procedural Skills (DOPS) tool is a tool to assess colonoscopic competency and includes ratings of the following domains: (i) assessment, consent and communication; (ii) safety and sedation; (iii) endoscopic skills during insertion and withdrawal; and, (iv) diagnostic and therapeutic ability. Scores range from 0-100, with higher scores representing higher colonoscopic competency. The tool will be used to assess participants during an integrated scenario. A change in these ratings before and after intervention is the secondary outcome.
Time Frame: 4-6 weeks after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Curriculum Group | Self-directed Learning Group
Number analyzed (Participants) | 16 | 17
units on a scale
  Colonoscopy-specific performance | 67 (12.1) | 54.3 (14.3)
  Communication skills | 83.1 (5.7) | 75.9 (9.7)
  Global performance | 69.4 (7) | 63.5 (8.8)

ADVERSE EVENTS:
Arm/Group | Curriculum Group | Self-directed Learning Group
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No